CLINICAL TRIAL: NCT01544647
Title: Comparison of 2 Spa Therapy Protocols in Symptomatic Knee Osteoarthritis : a Randomised Trial
Brief Title: Spa Therapy in Knee Osteoarthritis (OA): Nancy-thermal
Acronym: Nancythermal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-A01319-32
Record Dates: First submitted 2012-02-16; First posted 2012-03-06 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; spa therapy; spa modalities
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual spa protocol (Active Comparator): 4 treatments (massages, showers, mud and pool sessions) are provided 6 days a week during 3 weeks.
  Interventions: Other: Usual spa protocol
- Active spa protocol (Active Comparator): 4 treatments (massages, showers, mud and pool sessions) are provided 3 days a week during 3 weeks then patients will follow an exercise program 3 days a week during 3 week.
  Interventions: Other: Active spa protocol

INTERVENTIONS:
Other: Usual spa protocol — In the first group, 4 treatments (massages, showers, mud and pool sessions) are provided 6 days a week during 3 weeks.
  Arms: Usual spa protocol
Other: Active spa protocol — 4 treatments (massages, showers, mud and pool sessions) are provided 3 days a week during 3 weeks then patients will follow an exercise program 3 days a week during 3 week.
  Arms: Active spa protocol

SUMMARY:
Non-pharmacological treatments are recommended for the management of knee osteoarthritis (EULAR or OARSI recommendations) and some thermal modalities may be effective for relieving symptoms in knee Osteoarthritis. However supporting evidence is limited and nothing is known about the advantage of one modality of thermal therapy over another.

The main objective of the study is to compare the number of patients achieving a composite response criteria associating the minimal clinically important improvement at 6 months, defined as ≥ 19.9 mm on the visual analogue pain scale and/or ≥ 9.1 points in a normalised Western Ontario and McMaster Universities osteoarthritis index function score and no knee surgery in 2 spa therapy protocols (a "usual protocol" and an "active protocol") in knee osteoarthritis.

The secondary objectives are:

1. To compare the efficacy of the 2 protocols at 3 months.
2. To determine the evolution of quality of life and medical care consumption
3. To describe postural abnormalities
4. To determine predictive factors to a favourable response at 3 and 6 months

DETAILED DESCRIPTION:
This is a monocentric randomised non inferiority trial comparing 2 spa therapy protocols in symptomatic knee OA.

In the first group, 4 treatments (massages, showers, mud and pool sessions) are provided 6 days a week during 3 weeks. In the second group, the same 4 treatments are provided 3 days a week during 3 weeks then patients will follow an exercise program 3 days a week during 3 week.

Data will be collected at inclusion, 3 and 6 weeks and 3 and 6 months.

ELIGIBILITY:
Inclusion criteria are:

* both gender
* uni or bilateral symptomatic knee OA
* pain VAS > 3 on a 0-10 scale)
* fulfilling ACR criteria for knee OA
* Kellgren and Lawrence stage 2 or over on standard radiograph

Non inclusion criteria are:

* severe comorbidity
* isolated femoro-patellar knee OA
* total knee replacement surgery expected during the next year
* other joint disease
* a contraindication or intolerance to any aspect of spa treatment (immune deficiency, evolving cardiovascular conditions, cancer, infection),
* spa treatment within the previous 12 months
* knee injection within the past month for corticosteroids and within the past 3 months for hyaluronic acids
* osteoarthritis (SYSADOA) change in the past 3 months
* massages, physiotherapy or acupuncture in the past month
* Patients will not be allowed to modify their non-steroidal antiinflammatory drug (NSAID) or their analgesic drug within the past 5 days and in the previous 12 h respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Composite response criteria: achievement of the minimal clinically important improvement of pain VAS and/or the WOMAC score and no knee surgery | 6 months
  The main outcome endpoint is the number of patients achieving minimal clinically important improvement (MCII) at 6 months, defined as ≥19.9 mm on the visual analogue pain scale and/or ≥9.1 points in a normalised Western Ontario and McMaster Universities osteoarthritis index function score and no knee surgery.

SECONDARY OUTCOMES:
Achievement of the patient acceptable symptom state | 3 and 6 months
evolution of quality of life scores | 3 and 6 months
medical care consumption | 3 and 6 months
  particularly NSAIDs, pain killers
postural abnormalities | 3 and 6 months
  The method used aimed at evaluating two modalities of postural regulation - quiet stance and during movement - and their related neurosensory organization. Postural control during quiet stance will be evaluated with and without sensory conflict by a static posturographic test and by a sensory organization test; postural control during movement will be evaluated by a dynamic posturographic test with slow sinusoidal oscillations.
adverse events | 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy university hospital center, Nancy, France